CLINICAL TRIAL: NCT01369901
Title: Effect of Functional Exercise in Patients With Spinal and Bulbar Muscular Atrophy
Brief Title: Effect of Functional Exercise in Patients With Spinal Bulbar Muscular Atrophy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 110171; 11-N-0171
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-02-28

CONDITIONS: Motor Neuron Disease
Keywords: Exercise; Spinal Bulbar Muscular Atrophy; Spinal and Bulbar Muscular Atrophy; SBMA; Motor Neuron Disease
MeSH Terms: conditions — Motor Neuron Disease; Motor Activity; Bulbo-Spinal Atrophy, X-Linked

ARMS (2):
- Group A (Experimental): Functional exercise
  Interventions: Behavioral: A functional exercise program
- Group B (Active Comparator): Stretching exercise
  Interventions: Behavioral: A stretching exercise program

INTERVENTIONS:
Behavioral: A functional exercise program
  Arms: Group A
Behavioral: A stretching exercise program
  Arms: Group B

SUMMARY:
Background:

-Spinal and bulbar muscular atrophy (SBMA) is an inherited disorder that affects men. People with SBMA often have weakness throughout the body, including the muscles they use for swallowing, breathing, and speaking. We do not know if exercise helps or harms people with SBMA.

Objective:

-To see if a 12-week program of either functional exercise or stretching exercises will improve strength, function, or quality of life in people with SBMA

Eligibility:

* Participants will be men 18 years of age or older who have genetic confirmation of SBMA.
* They must be able to walk at least 50 feet with or without an assistive device such as a cane or a walker and stand for 10 minutes without using an assistive device.
* They must have access to a computer with an Internet connection.

Design:

* At the first visit to NIH (2 days), participants will have a medical history taken and undergo a physical exam. They will also have blood tests and an EKG, and complete questionnaires about mood, health, and exercise. Tests of muscle strength, balance, and endurance will also be done.
* Participants who qualify for the study will receive instruction about either strengthening or stretching exercises. They will do these exercises at home one to three times a week for 12 weeks.
* They will wear a small activity monitor while they exercise and record their exercise in a diary.
* At the end of 12 weeks, participants will return to the NIH for 2 days. They will undergo the same tests as they had on the first visit.
* Participants will receive follow-up phone calls and e-mails during the study and for 4 weeks after the last visit....

DETAILED DESCRIPTION:
Objective: Spinal and bulbar muscular atrophy (SBMA), or Kennedy s disease, is a slowly progressive, X-linked motor neuron disease for which there is currently no treatment. It is caused by a mutation in the androgen receptor that results in a polyglutamine repeat expansion. The role of exercise in motor neuron disease research is debated. Although SBMA is believed to be primarily a neuronopathy, the potential effect of aberrant androgen receptor activity on muscle leads exercise to be of uncertain utility in this population. Our objective is to examine the safety and efficacy of exercise regimens in Kennedy s disease.

Study Population: We aim to enroll 80 men with genetically confirmed Kennedy s disease.

Design: This will be a randomized, evaluator blinded, trial with 25 subjects in each exercise arm. Following informed consent, the subjects will undergo an initial medical and physical evaluations followed by a series of neurological tests and blood work over a two-day outpatient visit at the NIH. The subjects will provide blood work for analysis of hormonal levels and assessment of any potential muscle damage. On the second day of their visit, the subjects will be randomized and taught a series of either functional or stretching exercises that they will engage in as part of the study and control arms, respectively. Following the baseline visit to NIH, the subjects will be monitored throughout the study with telephone contacts and other measures including video recording to monitor their progress and compliance. The subjects will return to the NIH at the end of a 12 week period at which time the physical and laboratory testing will be repeated. After the 12 week exercise period there will be a four week period where we will follow-up with the participants by telephone and e-mail. At the end of the trial all of the subjects will be informed of the study results and given the opportunity to learn the exercises if they are found to be beneficial.

Outcome Measures: The primary outcome measure used will be the Adult Myopathy Assessment Tool (AMAT). Secondary outcome measures will involve quantitative muscle analysis (QMA), the Timed Up and Go (TUG) test, a quality of life measure (SF-36v2TM), adverse event questionnaires, a Computerized Dynamic Posturography (CDP) assessment of balance, accelerometer measurements of exercise effort, and progressive height sit-to-stand testing. Several exploratory biomarkers that may be affected by exercise will be evaluated, including insulin-like growth factor-1 (IGF-1), insulin-like growth factor binding protein 3, testosterone, growth hormone, and creatine kinase. Beck Depression Inventory (BDI) testing will also be used to determine if the subjects mood is affected by exercise. Qualitative sub-study questions, international index of erectile function, Block brief food questionnaire, Aggression Questionnaire, Activities-specific Balance Confidence (ABC) scale, Fatigue Symptom Inventory, and physical activity survey measures will also be employed.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Genetically confirmed SBMA.
  2. Ambulatory and walk a distance of at least 50 feet with or without a walker.
  3. Able to stand for 10 minutes without the use of any assistive devices.
  4. Willing to travel to the NIH at the beginning and end of the study.
  5. Willing to participate in telephone monitoring.
  6. AMAT score of less than 41, but greater than 14.
  7. Male.
  8. Willing to participate in all aspects of trial design and follow-up.
  9. Access to a computer with an internet connection
  10. Able to do all of the exercises according to the standards of the study examiners at the beginning and end of the study
  11. Willing to forgo starting an additional exercise plan for the 12 week duration of the study
  12. Age greater than 18 years

EXCLUSION CRITERIA:

1. Medical condition which would preclude exercise such as COPD, congestive heart failure, and cardiac arrhythmias.
2. Presence of an additional comorbid condition such as stroke, myopathy, or radiculopathy which also results in weakness.
3. Beginning a separate exercise program involving at least two weekly sessions of 20 minutes of exercise each within two months of the start of the trial.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-06-08; Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Adult Myopathy Assessment Tool (AMAT)

SECONDARY OUTCOMES:
To assess the effect of functional exercise on muscle strength as measured by quantitative muscle analysis (QMA), and the Timed up and go test (TUG), and progressive height sit-to-stand.
Several exploratory biomarkers that may be affected by exercise will be evaluated, including insulin-like growth factor-1 (IGF-1), testosterone, growth hormone, and creatine kinase.
To assess the ability of patients to maintain exercise compliance as measured by accelerometer measurements.
To assess the effect of functional exercise on balance as measured by Computerized Dynamic Posturography (CDP) evaluation.
To assess the effect of functional exercise on adverse outcomes as measured by an adverse event questionnaire.
Beck Depression Inventory (BDI) testing will also be used to determine if the subjects mood is affected by exercise.
To assess the effect of functional exercise on quality of life as measured by the SF36v2.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H Fischbeck, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kennedy WR, Alter M, Sung JH. Progressive proximal spinal and bulbar muscular atrophy of late onset. A sex-linked recessive trait. Neurology. 1968 Jul;18(7):671-80. doi: 10.1212/wnl.18.7.671. No abstract available. PMID 4233749
- [Background] Harding AE, Thomas PK, Baraitser M, Bradbury PG, Morgan-Hughes JA, Ponsford JR. X-linked recessive bulbospinal neuronopathy: a report of ten cases. J Neurol Neurosurg Psychiatry. 1982 Nov;45(11):1012-9. doi: 10.1136/jnnp.45.11.1012. PMID 6890989
- [Background] Olney RK, Aminoff MJ, So YT. Clinical and electrodiagnostic features of X-linked recessive bulbospinal neuronopathy. Neurology. 1991 Jun;41(6):823-8. doi: 10.1212/wnl.41.6.823. PMID 2046924